CLINICAL TRIAL: NCT04771299
Title: Efficacy of Cariprazine in Improving Cognitive Functioning in Euthymic Patients With Bipolar I Disorder: A Proof of Concept Randomized, Double Blind Placebo Controlled Trial
Brief Title: Assessing the Role of Cariprazine in Improving Cognition in Euthymic Bipolar Patients
Acronym: CARPZ-01
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Research support no longer available.
Sponsor: Lakshmi N Yatham (Other)
Responsible Party: Sponsor-Investigator, Lakshmi N Yatham, Investigator, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H20-01293
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Bipolar I Disorder; Cognitive Impairment
Keywords: Bipolar I Disorder; Euthymia; Cariprazine; Cognition; Memory
MeSH Terms: conditions — Cognitive Dysfunction | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cariprazine (Active Comparator): 1.5mg of Cariprazine added to their current treatment for 6 week period
  Interventions: Drug: Cariprazine
- Placebo (Placebo Comparator): Matching placebo added to their current treatment for 6 week period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cariprazine — Cariprazine is a novel atypical antipsychotic medication that has been approved by the Food and Drug Administration (FDA) for treatment of schizophrenia, manic or mixed, and depressive episodes associated with bipolar I disorder.
  Other Names: VRAYLAR®
  Arms: Cariprazine
Other: Placebo — Placebo is an inactive substance that looks identical to the study medication that contains no therapeutic ingredient.
  Arms: Placebo

SUMMARY:
Some patients with bipolar disorder show broad cognitive impairments (e.g. difficulty with concentration, problem solving, memory etc.) that persist during euthymia (no symptoms of depression or mania) despite remission of mood symptoms. Cognitive deficits (significant cognitive impairments) in bipolar disorder are associated with impairments in everyday functioning and quality of life. Thus, improving cognitive functioning is an important treatment goal in people with bipolar disorder. In a recent study, investigators have demonstrated that lurasidone; an atypical antipsychotic was more effective than treatment as usual in improving cognition. The study will examine the efficacy of Cariprazine (VRAYLAR®) in improving cognition in patients with bipolar disorder. Cariprazine is a novel atypical antipsychotic medication that has been approved by the Food and Drug Administration (FDA) for treatment of schizophrenia, manic or mixed, and depressive episodes associated with bipolar I disorder. This study is a randomized (like the flip of a coin), double-blind (participant and the study team will not know which treatment arm participant will receive) study in which 30 participants will be randomized across two sites in Canada.

DETAILED DESCRIPTION:
Specific Procedures: If participant agrees to take part in this study, the procedures and visits include the following:

Screening Visit: (approximately 3.0 hours):Prior to any procedures being conducted, the Informed Consent Form will be reviewed with participant in detail and participant will have the opportunity to decide if s/he wish to participate in the study or not. If participant meets all the requirements and all of participants questions have been answered, participant will be asked to sign the consent form. A clinical assessment will take place, where participant will be asked questions about participants medical and psychiatric history including family psychiatric history and prior treatments. Participants medical records may be reviewed to confirm diagnosis and treatment history. The study doctor will complete rating scales to determine the current status of participants mood. Participant may choose not to answer any questions that participant is uncomfortable with. Neurocognitive tests (i.e., paper and pencil tests of memory, problem solving etc. as well as a computer component) will be conducted to determine if cognitive impairment exists. If there is no cognitive impairment no further procedures will be conducted. The information that is collected from the participant will not be used for any purpose other than stating how many people were screened for study participation. If cognitive impairment does exist, participant will be scheduled to return to the clinic within 4 weeks and a baseline visit will be completed. In addition to the above procedures, participant will also have a physical examination, which includes measurement of participants height, weight and blood pressure. To ensure safety of participation in the study, participant will be asked to have routine clinical blood work, including a pregnancy test for female participants of childbearing age, and a urine test for a drug screen. If participant has a personal or family history of significant cardiac problems or show cardiac abnormalities on the physical exam an EKG will be performed.

Baseline Visit (approximately 3-3.5 hours): At baseline, rating scales and clinical assessment will be completed to determine the current status of participants mood. Information about participants current medications and any side effects will be obtained. If participant is not eligible, participants will not be randomized into the study and no further procedures will be conducted.

If participant is eligible, participant will be randomized to receive either cariprazine or placebo in addition to participants current medications, and instructed on dosing. Participant will complete more neurocognitive testings. The use of benzodiazepines (Ativan, Lorazepam etc.) within 4 hours or caffeine intake 2 hours prior to neurocognitive testing is not allowed. Participant will be asked to complete questionnaires about participants functioning and quality of life. Vital signs and weight measurements will be obtained. Study medication will be dispensed to last until the next clinic visit. Participant must bring the remaining unused medication to the next appointment. Participant is asked to give 1.5 tablespoons (20 ml) of blood to analyze markers which may be predictive of bipolar disorder (biomarkers). Biomarkers are substances (like proteins, protein particles, or chemicals that make body function) that may be altered in those with bipolar disorder or may provide information about treatment response. These samples will be labelled with a unique study number and will not contain any identifying information. The samples will be stored at the study site until they are sent for analysis at the end of the study.

Weeks 1, 2 and 4: (approximately 15 minutes each): Participant will be contacted by telephone to review any changes to participants medications and any side effects that may be experienced.

Week 3 Clinic appointment: (approximately 1 hour) : A clinical assessment will take place, where participant is asked questions about their mood. Information about participants current medications and any side effects will be obtained. Vital signs and weight measurements will be obtained. Bottle-1 of the study medication will be collected and bottle-2 of study medication will be dispensed. Participant will be asked to bring the remaining unused study medication from bottle-2 to the next clinic appointment. Participant will be asked to give a tablespoon (15 ml) of blood to test for levels of study medication. The samples will be labelled with a unique study number and will not contain any identifying information. The samples will be stored at study site until they are sent for analysis at the end of the study.

Week 6/ Early Termination Visit: (approximately 3 hours): A clinical assessment will take place where participant will be asked questions about their mood. Neurocognitive testing will be administered to all participants who have had a minimum of 3 weeks of double- blind treatment. Participant is asked to complete some questionnaires about participants functioning and quality of life. Information about participants current medications and any side effects will be obtained. Vital signs and weight measurements will be obtained. Participant will have a physical examination and will be asked to complete routine laboratory tests including a pregnancy test for female participants of childbearing age, and a urine drug screen. In addition, participant is asked to give 2 tablespoons (30 ml) of blood to measure levels of study medication, and biomarkers. These samples will be labelled with a unique study number and will not contain any identifying information. The samples will be stored at study site until they are sent for analysis at the end of the study.

Follow-up Telephone Assessment (2 weeks after study completion; approximately 15 minutes): Participant will be contacted by telephone to assess any side effects or issues post treatment.

ELIGIBILITY:
Participant Inclusion Criteria Participants who meet all of the following criteria are eligible to participate in this trial.

1. Males or females aged 19 to 65 years inclusive.
2. DSM-5 diagnosis of Bipolar I Disorder, with or without a history of psychosis.
3. All patients must be taking either a mood stabilizer (i.e. lithium or valproate) or an atypical antipsychotic, or a combination of these (two mood stabilizers or a mood stabilizer plus an atypical antipsychotic), at therapeutic doses, for mood stabilization. Those taking two or more atypical antipsychotics are excluded. Medications and therapeutic doses are: lithium, serum level 0.6-1.2 mEq/L; divalproex/sodium valproate, serum level 350-700 mM/L (45-125 mcg/ml); risperidone 1-6 mg/day; olanzapine 5-20 mg/day; quetiapine IR or XR 300-800 mg/day; aripiprazole 10-30 mg/day; asenapine 5-20 mg/day, or ziprasidone 80-160 mg/day.
4. All concomitant medication must be at a stable dose for a minimum of two weeks prior to randomization.
5. Clinically stable during the last 4 weeks, as assessed by clinical interview, prior to the randomization visit.
6. A MADRS and YMRS score less than or equal to 8.
7. Patients who show cognitive impairments, defined as 0.5 standard deviations below the mean or worse (Z = -0.5 or lower), on either the WAIS-IV Coding subtest, or the RAVLT total learning score on trials 1-5 or immediate recall trial, at screening visit.
8. A WAIS-IV vocabulary scaled score ≥ 5 (equivalent to estimated IQ 80 or greater).
9. A sufficient level of English language.
10. Females who are postmenopausal for at least 1 year before the screening visit (confirmed by an FSH test) or are surgically sterile.
11. Females of childbearing potential who are taking contraceptive pills or agree to practice highly effective double barrier methods of contraception, from the time of signing the informed consent up to the last dose of study drug, and for 7 days after the last dose. Abstinence will only be considered an adequate form of contraception if it is the usual and preferred method.
12. Capability of understanding, consenting to, and complying with study requirements, study visits, and to return to the clinic for follow-up evaluations as specified by the protocol.

4.2 Participant Exclusion Criteria Participants meeting any of the following criteria are not eligible to participate in the trial.

1. A history of unstable or inadequately treated medical illnesses including moderate to severe brain injury, or neurological illnesses impacting cognitive function. Patients with a personal or family history of cardiac problems will need to undergo EKG at screen visit, and will be excluded if results are abnormal.
2. Participants taking procognitive medications, clozapine, tricyclic antidepressants, first-generation antipsychotics, benztropine, cogentin or lurasidone at screening visit.
3. Those taking two or more antipsychotics.
4. Anticholinergics and stimulants that increase dopamine levels are not permitted.
5. Cognitive remediation therapy within 3 months prior to entry or during the double blind phase.
6. Neuromodulation treatment with ECT or DBS within 8 weeks, or rTMS, tDCS or experimental drug treatment within 30days.
7. History of nonresponse or intolerance to cariprazine.
8. Psychiatric disorder other than bipolar disorder.
9. Participants who currently meet criteria for anxiety disorder (GAD, OCD, panic disorder, PTSD).
10. Those with a current or lifetime diagnosis of ADHD or other learning disorders.
11. Those meeting DSM-5 criteria for alcohol or substance abuse or dependence disorder within the past month.
12. Significant risk of harm to self or others.
13. Those with severe personality disorders causing significant impairment in functioning.
14. Pregnancy or lactation.
15. Liver function tests (AST and ALT) three times the upper limit of normal.
16. Contraindications to cariprazine according to prescribing information.
17. Participants with increased risk or diagnosis of impulsive or compulsive behavior

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-09-08 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
Improvement in cognitive performance | 6 weeks
  The primary efficacy measure will be improvement in cognitive performance, as measured by changes in composite cognitive score from baseline to endpoint, extracted from the International Society for Bipolar Disorders-Battery for Assessment of Neurocognition. The higher the scores the better the outcome.
Improvement in functioning | 6 weeks
  The co-primary efficacy measure will include changes in functioning from baseline to endpoint measured using UCSD based performance skills assessment-brief version. The higher the scores the better the outcome.

SECONDARY OUTCOMES:
Change in depression | 6 weeks
  Montgomery Asberg Depression Rating Scale will be used to assess changes in bipolar depression from baseline to endpoint. Lower scores reflect better clinical outcomes.
Change in Mania | 6 weeks
  The Young Mania Rating Scale will be used to assess changes in mania from baseline to endpoint. The higher the scores means worsening in Mania. Lower scores reflect better clinical outcomes.
Improvement in overall psychiatric status | 6 weeks
  Clinical Global Improvement Scale will be used to assess change from baseline to endpoint in overall psychiatric status. The higher the scores means worsening in psychiatric status .
Improvement in Quality of Life | 6 weeks
  Quality of Life, Bipolar Version Scale will be used to assess improvement in quality of life from baseline to endpoint. Higher scores reflect better outcomes.
Improvement in Subjective-rated Cognitive Functioning | 6 weeks
  Cognitive Complaints in Bipolar Disorder Rating Assessment will be used to assess changes in subjective cognitive functioning from baseline to endpoint. Lower scores mean better outcomes.
Improvement in Objectively Rated Daily Functioning | 6 weeks
  Functioning Assessment Short Test will be used to assess improvement in objectively rated daily functioning, defined as change in scores from baseline to endpoint. Higher scores mean better outcomes.
Improvement in Subjectively Rated Daily Functioning | 6 weeks
  Sheehan Disability Scale (SDS) will be used to assess improvement in subjectively rated daily functioning, defined as change in scores from baseline to endpoint. Lower scores mean better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi N Yatham, MBBS,MRCPsyc, Principal Investigator — University of British Columbia, Department of Psychiatry, BC
Locations (1):
- Djavad Mowfaghian Centre for Brain Heath, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No